CLINICAL TRIAL: NCT04185610
Title: IIT2019-07-ASHER-QIGONG: A Mind-Body Intervention for Chemotherapy-Induced Peripheral Neuropathy
Brief Title: A Mind-Body Intervention for Chemotherapy-Induced Peripheral Neuropathy
Acronym: QiGong
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: Arash Asher, MD (Other)
Responsible Party: Sponsor-Investigator, Arash Asher, MD, Director, Cancer Rehabilitation & Survivorship, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2019-07-ASHER-QIGONG
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Cancer
Keywords: Qi Gong
MeSH Terms: conditions — Neoplasms | interventions — Qigong

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Qi Gong (Experimental): Weekly QiGong for Chemotherapy-Induced Neuropathy classes for 10 weeks
  Interventions: Other: Qi Gong

INTERVENTIONS:
Other: Qi Gong — Guided Qi Gong class

SUMMARY:
This pilot study will include up to 25 patients with cancer experiencing chemotherapy-induced peripheral neuropathy. Patients enrolled in the study will participate in a 10-week QiGong for Chemotherapy-Induced Neuropathy program. Patients will be evaluated before and after their program participation. Within 2 weeks before the program start date, patients will be administered an objective neuropathy assessment by a physician or nurse, and will complete questionnaires assessing chemotherapy-induced peripheral neuropathy, perceived cognitive functioning, quality of life, and cancer-related symptoms. Patients will repeat these assessments at the end of the last QiGong class and will be asked to provide feedback on the QiGong program as a whole. Self-report questionnaires will also be repeated one week after the last class.

Total duration of subject participation will be 11-13 weeks. Total duration of the study is expected to be approximately 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer, stage 1-4.
* Completed taxane- or platinum-based chemotherapy at least three months (90 days) ago but within 24 months of signing consent. Current use of anti-estrogen therapy, Herceptin, or PARP inhibitors is okay.
* Experiencing at least grade 1 peripheral sensory neuropathy, peripheral motor neuropathy, or dysesthesias based on the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4 (NCI CTCAE v4.0).
* Age ≥ 18 years.
* Concomitant use of analgesics is permitted if the dose has been stable for at least 2 weeks prior to study enrollment (no new analgesics have been added, discontinued, or changed in the 2 weeks prior to study enrollment).
* Reasonable functional stability as assessed by the evaluating physician.
* Must be able to understand and communicate proficiently in English.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Syphilis, alcoholic neuropathy, diabetic neuropathy, neurological disorders, brain injury, or stroke, as assessed by the treating physician.
* Medical history of neuropathy from any type of nerve compression (e.g., carpal tunnel or tarsal tunnel syndrome, radiculopathy, spinal stenosis, brachial plexopathy, leptomeningeal carcinomatosis), as assessed by the treating physician.
* Neuropathy related to abnormal TSH or B12 levels as assessed by treating physician
* Current severe depression, suicidal ideation, bipolar disease, alcohol abuse, or major eating disorder, as assessed by the treating physician.
* Severe personality disorder or psychiatric disorder that would interfere with participation in a QiGong program, as assessed by the evaluating physician.
* Currently participating in another QiGong or Tai Chi program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Objective Modified Total Neuropathy Scale (mTNS) score | 10 weeks
  Change in the Modified Total Neuropathy Scale (mTNS) score from Baseline to T1 (last day of class)
Subjective Neurotoxicity Subscale score | 11 weeks
  Change in the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity (FACT/GOG-NTX) Subscale Score from Baseline to T1 (last day of class) and T2 (1-week follow-up).

SECONDARY OUTCOMES:
Attendance | 10 weeks
  Number of QiGong classes attended by those who enroll
Retention | 10 weeks
  Completion of both pre- and post-assessments
Patient Interest | 1 week
  Percentage of patients approached who sign consent
Patient Evaluation of QiGong Program | 1 day
  Scores on the evaluation titled: QiGong Program Evaluation. Study participants will provide a score for 3 questions related to the QiGong intervention. The minimum value is 0 and maximum value is 4, and higher score means a better outcome.
  Participants will also be asked 4 additional questions about the class. The minimum value is 0 and the maximum value is 10, and higher score means a better outcome.
  A composite of all the scores for each participant will be calculated, with higher scores indicating a better outcome.
Perceived cognitive functioning | 11 weeks
  Change in the Functional Assessment of Cancer Therapy - Cognition (FACT-Cog) score from Baseline to T1 (last day of class) and T2 (1-week follow-up).
Physical Well-Being | 11 weeks
  Change in the FACT/GOG-NTX Physical Well-Being Subscale Score from Baseline to T1 (last day of class) and T2 (1-week follow-up).
Social/Family Well-Being | 11 weeks
  Change in the FACT/GOG-NTX Social/Family Well-Being Subscale Score from Baseline to T1 (last day of class) and T2 (1-week follow-up).
Emotional Well-Being | 11 weeks
  Change in the FACT/GOG-NTX Emotional Well-Being Subscale Score from Baseline to T1 (last day of class) and T2 (1-week follow-up).
Functional Well-Being | 11 weeks
  Change in the FACT/GOG-NTX Functional Well-Being Subscale Score from Baseline to T1 (last day of class) and T2 (1-week follow-up).
Impact on symptom experience | 11 weeks
  Change in the ESAS scores from Baseline to T1 (last day of class) and T2 (1-week follow-up).

CONTACTS AND LOCATIONS:
Overall Officials: Arash Asher, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States